CLINICAL TRIAL: NCT04268433
Title: Musical Heart Rhythm Regulation: The MUSIC-HR Study
Brief Title: The MUSIC-HR Study
Status: Completed | Type: Observational
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Collaborators: CW+ Charity (Other)
Responsible Party: Sponsor
Other Study IDs: C&W18/005; 242951 (Other: Integrated Research Application System)
Record Dates: First submitted 2020-02-10; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Musical Heart Rhythm Regulation; Cardiovascular Diseases; Heart Rate Control
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: N/A - Non-interventional study — Stages:
  1. Patient information and written informed consent (3 Copies. To be carried out >24 hours after receiving the patient information sheet)
  2. Physiological recording set up (ECG, BP, sensor and respiratory band)
  3. Control period - no music played
  4. Series of pieces of music without tempo control
  5. Repeat series of pieces of music with tempo control
  6. Participant leaves the study

SUMMARY:
The idea that music has an effect on heart rate and blood pressure has existed for some time. In 1918, Hyde and Scalapino [1] reported that minor tones increased pulse rate and lowered blood pressure, whereas "stirring" music increased both blood pressure and heart rate. In the management of many cardiovascular disorders heart rate control is paramount. Furthermore, many cardiovascular investigations (e.g. Cardiac CT) require adequate heart rate control in order to achieve diagnostic images and therefore results. Whilst pharmacologic therapy is available and remains the main strategy for heart rate control, this is not always without consequences. Side effect profiles, patient intolerance and also variable efficacy are limiting factors for pharmacological therapy. Alternative strategies to achieve adequate heart rate control are therefore needed.

The aim of this study is to explore the potential use of music to control heart rates and other physiological parameters such as respiratory rate and blood pressure. The central study team hypothesize that by changing the tempo of the music they will be able to influence the natural variations in heart rate.

1. Hyde IM, Scalapino W. The influence of music upon electrocardiograms and blood pressure. Am J Physiol.1918;46:35-38.

DETAILED DESCRIPTION:
This is a single-arm non-randomized pilot study. Staff at Chelsea and Westminster NHS Foundation Trust will be recruited via the placement of posters in staff only areas such as staff rooms and via the daily communications that the Trust use. Those who meet all of the inclusion criteria and none of the exclusion criteria will be approached for participation in the study. The participants will be asked to listen to a series of musical genres, selected in random order, whilst lying on a standard hospital bed for comfort. This will take place in a private clinical room to minimise disturbance and any variation in heart rate caused by external stressors. The participants will have an ECG recording performed by attachment of adhesive surface lead electrodes to the chest and arms. This will be continuous throughout the protocol. They will also have a continuous non-invasive blood pressure recording using equipment that is in routine clinical practice (Finapress BP) and respiration monitored via a respiration belt. They will also be asked to wear a small lightweight sensor that gives readings of heart rate and blood pressure at 2 minute intervals.

After a period of approximately 10 minutes of ECG recording without music (control period), a series of pieces of music will be played whilst the ECG recordings continue. Each piece of music will last for no more than 5 minutes, 3 will be selected by the investigators and one will be pre-chosen by the participant prior to their attendance. The order in which these pieces will be played will be chosen at random. There will be a 3 minute recovery time in between each piece of music. The same pieces of music will then be played back to the participant but this time the music will subtly change tempo in reaction to the patient's heart rate. This is achieved by the ECG feeding data into the computer playing the music, whereupon the data is processed by Max MSP software and used to control the playback speed in Ableton Live. The algorithm for change is a linear one: the higher a patient's heart rate is in relation to a desired bpm target, the more the music will slow down. (There will be a limit to the extent of the tempo adjustment, in order to prevent any noticeable distortion to the music.)

The tempo of the music is controlled by computer. The ECG recording will feed into the computer where the software alters the tempo of the music based on the real-time heart rate feedback. The hypothesis is that by altering the tempo of the music the investigators will see changes in the heart rate of the participant. These changes will then feedback to the software which will continue to alter the tempo accordingly with the aim to achieve a degree of heart rate control and see less heart rate variation and less high heart rates. It should take around one hour to complete all the study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Employed by Chelsea and Westminster NHS Foundation Trust with any contract type (substantive, fixed term, honorary or bank)
* Age 18 or above
* Capable of giving informed consent
* Normal 12 lead ECG and blood pressure recording

Exclusion Criteria:

* Under 18 years of age
* Incapable of giving informed consent
* Regular use of any medications that interact with physiological control of the parameters being measured
* Hearing impairment
* Skin sensitivity to ECG electrodes

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: As above.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of the effect of music and music tempo on heart rate control | Participants will be involved in the study for a total of 1 day. No follow-up is required so data will be ready for analysis after participants have completed the music exercise.
  After a period of approximately 10 minutes of ECG recording without music (control period), a series of pieces of music will be played whilst the ECG recordings continue. Each piece of music will last for no more than 5 minutes, 3 will be selected by the investigators and one will be pre-chosen by the participant prior to their attendance. The order in which these pieces will be played will be chosen at random. There will be a 3 minute recovery time in between each piece of music. The same pieces of music will then be played back to the participant but this time the music will subtly change tempo in reaction to the patient's heart rate. This is achieved by the ECG feeding data into the computer playing the music, whereupon the data is processed by Max MSP software and used to control the playback speed in Ableton Live. The algorithm for change is a linear one: the higher a patient's heart rate is in relation to a desired bpm target, the more the music will slow down.

SECONDARY OUTCOMES:
Assessment of the effect of music and music tempo on blood pressure and variability | Participants will be involved in the study for a total of 1 day. No follow-up is required so data will be ready for analysis after participants have completed the music exercise.
  As well as having an ECG recording performed, participants will also have a continuous non-invasive blood pressure recording using equipment that is in routine clinical practice (Finapress BP) and respiration monitored via a respiration belt. They will also be asked to wear a small lightweight sensor that gives readings of heart rate and blood pressure at 2 minute intervals.
  The data obtained from all of the physiological recordings with be analysed for associations.
Assessment of the effect of music on heart rate variability | Participants will be involved in the study for a total of 1 day. No follow-up is required so data will be ready for analysis after participants have completed the music exercise.
  As well as having an ECG recording performed, participants will also have a continuous non-invasive blood pressure recording using equipment that is in routine clinical practice (Finapress BP) and respiration monitored via a respiration belt. They will also be asked to wear a small lightweight sensor that gives readings of heart rate and blood pressure at 2 minute intervals.
  The data obtained from all of the physiological recordings with be analysed for associations.
Assessment of the effect of music on markers of repolarization instability | Participants will be involved in the study for a total of 1 day. No follow-up is required so data will be ready for analysis after participants have completed the music exercise.
  Effect of music on markers of repolarization instability (QT interval and T wave vector assessment).
Effect of music on cardiac autonomics | Participants will be involved in the study for a total of 1 day. No follow-up is required so data will be ready for analysis after participants have completed the music exercise.
  This is assessed by frequency analysis of ECG.
Assessment of the effect of music and music tempo on respiratory rate and variability | Participants will be involved in the study for a total of 1 day. No follow-up is required so data will be ready for analysis after participants have completed the music exercise.
  Respiration of participants will be monitored via a respiration belt whilst they are listening to music.

CONTACTS AND LOCATIONS:
Overall Officials: Sadia Khan, Principal Investigator — Chelsea and Westminster NHS Foundation Trust
Locations (1):
- Chelsea and Westminster Hospital, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hyde IM, Scalapino W. The influence of music upon electrocardiograms and blood pressure. Am J Physiol. 1918;46:35-38.